CLINICAL TRIAL: NCT03878667
Title: Effects of Calcium Supplementation on Body Composition, Metabolism and Exercise Capacity in Post-Menopausal Women Participating in the Curves for Women Fitness and Weight Loss Program
Brief Title: Effects of Calcium Supplementation on Women in the Curves for Women Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Richard B. Kreider, Executive Director, Human Clinical Research Facility, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2008-0643
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Diet Modification
Keywords: Calcium Supplementation; Exercise Intervention
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Diet (Placebo Comparator): No diet or exercise or calcium intervention
  Interventions: Dietary Supplement: Curves Calcium; Dietary Supplement: Calcium Carbonate; Dietary Supplement: Placebo
- High Calorie Diet (Experimental): High calorie (2,600 calorie) diet and exercise and calcium
  Interventions: Dietary Supplement: Curves Calcium; Dietary Supplement: Calcium Carbonate; Dietary Supplement: Placebo
- Low Carbohydrate/High Protein Diet (Experimental): Low carbohydrate (63% protein, 7% carbohydrate, 30% fat) diet and exercise and calcium
  Interventions: Dietary Supplement: Curves Calcium; Dietary Supplement: Calcium Carbonate; Dietary Supplement: Placebo
- High Carbohydrate/Low Protein (Experimental): High carbohydrate (15% protein, 55% carbohydrate, 30% fat) diet and exercise and calcium
  Interventions: Dietary Supplement: Curves Calcium; Dietary Supplement: Calcium Carbonate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curves Calcium — Curves Essential Bio-Available Calcium (providing 800 mg/d of calcium [as calcium citrate malate and calcium citrate], 400 IU/d of Vitamin D, 300 mg/d of magnesium, 4 mg/d of zinc, 2 mg/d of copper, 2 mg/d of manganese, 198 mg/d of potassium, 100 mg/d of trace mineral complex, and 2 mg/d of boron).
Dietary Supplement: Calcium Carbonate — Calcium (providing 950 mg/d as carbonate)
Dietary Supplement: Placebo — Dextrose placebo

SUMMARY:
The purpose of this study is to examine the effects of dietary calcium supplementation on weight loss, bone density, and markers of health and fitness in women participating in the Curves exercise and diet program.

DETAILED DESCRIPTION:
The Curves International fitness and weight loss program has become a very popular means of promoting health and fitness among women. The program involves a 30-minute circuit training program and a weight management program involving periods of moderate caloric restriction (1,200 to 1,600 calories per day) followed by short periods of higher caloric intake (2,600 calories per day). The program is designed to promote a gradual reduction in body fat while increasing strength and muscle mass/tone. Researchers in the Exercise & Sport Nutrition Lab at Texas A&M University have conducted an extensive study on the effectiveness and safety of the Curves fitness and diet program. Results of this initial study have shown that the program promotes weight loss, improves markers of health, and improves fitness. However, we feel that the program may be even more effective with some additional nutritional interventions. Calcium has been shown to slow bone loss and more recently has been found to help promote fat loss. If this is the case, supplementing the diet with calcium may promote greater benefits in women participating in the Curves fitness/diet program. The purpose of this study is to examine the effect of dietary calcium supplementation on weight loss, bone density, and markers of health and fitness in women participating in the Curves exercise and diet program.

ELIGIBILITY:
Inclusion Criteria:

* Participant is female;
* Participant is post-menopausal;
* Participant is between the ages of 45 and 65;
* Participant is sedentary, overweight (BMI > 27) and post-menopausal;

Exclusion Criteria:

* Participant has any metabolic disorder including known electrolyte abnormalities, heart disease, arrhythmias, diabetes, or thyroid disease;
* Participant has a history of hypertension, hepatorenal, musculoskeletal, autoimmune or neurological disease;
* Participant is taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive or androgenic medications;
* Participant has taken ergogenic levels of nutritional supplements that may affect muscle mass (i.g., creatine, HMB, etc.), anabolic/catabolic hormone levels (i.e., androstenedione, DHEA, etc.) or weight loss (i.e., ephedra, thermogenics, etc.) within three months prior to the start of the study;
* Participant is consistently taking 500 mg or more of a Calcium supplement per day;
* Participant is receiving Hormone Replacement Therapy (HRT);
* Participant is involved in a planned exercise program within 3 - 6 months prior to the start of the study;
* Participant has lost > 20 lbs. within the last 3 - 6 months;

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2005-12-31 (Actual)

PRIMARY OUTCOMES:
Body Composition: Body Fat | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in body composition (% body fat) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Fat Free Mass | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in body composition (fat free mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Bone Mass | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in body composition (bone mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Fat Mass | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in body composition (fat mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Lean Mass | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in body composition (lean mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Body Weight | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in body weight (lbs. body weight) obtained via digital scale and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Energy Homeostasis: Resting Energy Expenditure (REE) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in REE obtained via metabolic cart and expressed in absolute (kcals/d) and relative terms (kcals/kg/d) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's)
Energy Homeostasis: Respiratory Exchange Ratio (RER) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in RER as an indicator of carbohydrate and fat oxidation analyzed with related resting energy expenditure outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean changes from baseline with 95% confidence intervals (CI's)

SECONDARY OUTCOMES:
Muscular Strength: 1 Repetition Maximum (1RM) Bench Press | Measured prior to supplementation (Pre), after 10 weeks and 14 weeks
  Changes in bench press 1RM obtained from a bench press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Strength: 1 Repetition Maximum (1RM) Leg Press | Measured prior to supplementation (Pre), after 10 weeks and 14 weeks
  Changes in leg press 1RM obtained from a leg press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Endurance: 80% of 1 Repetition Maximum (1RM) Bench Press Endurance Test | Measured prior to supplementation (Pre), after 10 weeks and 14 weeks
  Changes in total repetitions at 80% of 1RM obtained from a bench press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Endurance: 80% of 1 Repetition Maximum (1RM) Leg Press Endurance Test | Measured prior to supplementation (Pre), after 10 weeks and 14 weeks
  Changes in total repetitions at 80% of 1RM obtained from a leg press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Body Water | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in body water obtained via Bioelectrical Impedance Analysis (BIA) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: Cholesterol | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: HDL Cholesterol | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in HDL cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: LDL Cholesterol | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in LDL cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: Triglycerides | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in triglycerides obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Glucose | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in glucose obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Calcium | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in calcium obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Albumin | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in albumin obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Total Protein | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in total protein obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Sodium | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in sodium obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Potassium | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in potassium obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Carbon Dioxide (CO2) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in carbon dioxide (CO2) obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Chloride | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in chloride obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Blood Urea Nitrogen (BUN) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in blood urea nitrogen (BUN) obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Creatinine | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in creatinine obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Alkaline Phosphatase (ALP) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in alkaline phosphatase (ALP) obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Amino Transferase (ALT) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in alanine amino transferase (ALT) obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Amino Transferase (AST) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in alanine amino transferase (ALT) obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel - CMP: Bilirubin | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in bilirubin obtained via venous blood draws (comprehensive metabolic panel - CMP) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: White Blood Cell (WBC) Count | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in white blood cell count (WBC) obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: White Blood Cell Differential | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in white blood cell differential obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Red Blood Cell (RBC) Count | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in red blood cell count obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Red Cell Distribution Width (RDW) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in red cell distribution width (RDW) obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Hemoglobin | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in hemoglobin obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Hematocrit | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in hematocrit obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Platelet Count | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in platelet count obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Mean Platelet Volume (MPV) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in mean platelet volume (MPV) obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Neutrophils | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in neutrophils obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Lymphocytes | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in lymphocytes obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Basophils | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in basophils obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Eosinophils | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in eosinophils obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Monocytes | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in monocytes obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Mean Corpuscular Volume (MCV) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in mean corpuscular volume (MCV) obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Mean Corpuscular Hemoglobin (MCH) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in mean corpuscular hemoglobin (MCH) obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Complete Blood Count - CBC: Mean Corpuscular Hemoglobin Concentration (MCHC) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in mean corpuscular hemoglobin concentration (MCHC) obtained via venous blood draws (complete blood count - CBC) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hormones: Insulin | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in serum insulin obtained from venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hormones: Leptin | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in serum leptin obtained from venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Heart Rate (HR) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in resting heart rate (HR) obtained via a blood pressure meter and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Systolic Blood Pressure (SBP) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in resting systolic blood pressure (mmHg) analyzed with related resting hemodynamic outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Diastolic Blood Pressure (DBP) | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in resting diastolic blood pressure (mmHg) analyzed with related resting hemodynamic outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Waist Circumference | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in waist circumference obtained via tape measure and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Hip Circumference | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in hip circumference obtained via tape measure and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Waist to Hip Ratio | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in the ratio of waist to hip (waist/hip circumference) analyzed with related anthropometric outcomes measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Body Mass Index | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in body mass index (kg of body mass/height in meters squared) analyzed with related anthropometric outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Cardiac Variable: Resting Electrocardiogram (ECG) | Measured prior to supplementation (Pre), after 10 weeks and 14 weeks
  Changes in resting ECG obtained via electrodes and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Exercise Capacity: Graded Exercise Test (GXT) | Measured prior to supplementation (Pre), after 10 weeks and 14 weeks
  Changes in exercise capacity obtained via a treadmill test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Subjective Rating of Quality of Life | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Changes in Quality of Life (QOL) obtained via SF36v2 questionnaire and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's). The SF-36 QOL inventory provides scores that assess physical functioning (i.e., ability to perform most vigorous physical activities without limitation to health); role physical (i.e., ability to work and perform daily activities); bodily pain (i.e., limitations due to pain); general health (i.e., assessment of personal health); vitality (i.e., feelings of energy); social functioning (i.e., ability to perform normal social activities); role emotion (i.e., problems with work or other daily activities); and, mental health (state of feelings of peacefulness, happiness, and calm) domains on a 0 (low) to 100 (high scale.
Subjective Rating of Appetite | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of appetite using the following scale: 0 (none), 1 - 3 (low), 4 - 6 (moderate), 7 - 9 (high), 10 (severe). Data will be analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Subjective Rating of Hunger | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of hunger using the following scale: 0 (none), 1 - 3 (low), 4 - 6 (moderate), 7 - 9 (high), 10 (severe). Data will be analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Subjective Rating of Satisfaction from Food | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of satisfaction from food using the following scale: 0 (none), 1 - 3 (low), 4 - 6 (moderate), 7 - 9 (high), 10 (severe). Data will be analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Subjective Rating of Feelings of Fullness | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of feelings of fullness using the following scale: 0 (none), 1 - 3 (low), 4 - 6 (moderate), 7 - 9 (high), 10 (severe). Data will be analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Subjective Rating of Amount of Energy | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of amount of energy using the following scale: 0 (none), 1 - 3 (low), 4 - 6 (moderate), 7 - 9 (high), 10 (severe). Data will be analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Subjective Rating of Overall Quality of Diet | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  A subjective Likert scale that asked participants to rank the frequency and severity of their symptoms of overall quality of diet using the following scale: 0 (none), 1 - 3 (low), 4 - 6 (moderate), 7 - 9 (high), 10 (severe). Data will be analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Dietary Energy Intake - Total Caloric Intake | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in caloric/energy intake (kcals/day) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Dietary Energy Intake - Carbohydrate | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in dietary carbohydrate intake (grams/day and grams/kg/day) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Dietary Energy Intake - Fat | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in dietary fat intake (grams/day and grams/kg/day) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Dietary Energy Intake - Protein | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in dietary protein intake (grams/day and grams/kg/day) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Perceptions of Side Effects - Dizziness | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in perceptions of dizziness using a Likert scale [0 (none), 1 - 4 (light), 5 - 6 (mild), 7 - 9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Perceptions of Side Effects - Headache | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in perceptions of headache using a Likert scale [0 (none), 1 - 4 (light), 5 - 6 (mild), 7 - 9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Perceptions of Side Effects - Tachycardia | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in perceptions of tachycardia using a Likert scale [0 (none), 1 - 4 (light), 5 - 6 (mild), 7 - 9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Perceptions of Side Effects - Palpitations | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in perceptions of palpitations using a Likert scale [0 (none), 1 - 4 (light), 5 - 6 (mild), 7 - 9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Perceptions of Side Effects - Dyspnea | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in perceptions of dyspnea using a Likert scale [0 (none), 1 - 4 (light), 5 - 6 (mild), 7 - 9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Perceptions of Side Effects - Nervousness | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in perceptions of nervousness using a Likert scale [0 (none), 1 - 4 (light), 5 - 6 (mild), 7 - 9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Perceptions of Side Effects - Blurred Vision | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in perceptions of blurred vision using a Likert scale [0 (none), 1 - 4 (light), 5 - 6 (mild), 7 - 9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Perceptions of Side Effects - Other Side Effects | Measured prior to supplementation (Pre), after 2 weeks, 10 weeks, 11 weeks and 14 weeks
  Change in perceptions of other side effects using a Likert scale [0 (none), 1 - 4 (light), 5 - 6 (mild), 7 - 9 (severe), or 10 (very severe)] and analyzed with related side effect outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No